CLINICAL TRIAL: NCT02166710
Title: Effect of Adductor Canal Femoral Nerve Block Compared to a Simulated Block on Knee Extensor Muscle Strength Following Total Knee Arthroplasty
Brief Title: Effect of Adductor Canal Nerve Block Compared to a Simulated Block on Quadriceps Strength Following Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14.093
Record Dates: First submitted 2014-06-05; First posted 2014-06-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Knee Arthroplasty
Keywords: Knee arthroplasty; Adductor canal block; Quadriceps strength

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor canal femoral nerve blockade (Experimental): Patients will receive continuous adductor canal femoral nerve blockade for 48 hours with a catheter connected to a pump infusing bupivacaine 0.125% and multi-modal analgesia for pain management following total knee arthroplasty. Knee extensor muscle strength will be measured at different time-points prior and after surgery.
  Interventions: Device: Adductor canal femoral nerve block
- Simulated nerve blockade (Placebo Comparator): Patients will receive a simulated continuous femoral nerve block at the level of the adductor canal for 48 hours with a catheter connected to a pump infusing bupivacaine 0.125% and multi-modal analgesia for pain management following total knee arthroplasty. Knee extensor muscle strength will be measured at different time-points prior and after surgery.
  Interventions: Device: Simulated nerve blockade

INTERVENTIONS:
Device: Adductor canal femoral nerve block — A 18 Gauge Tuohy needle will be inserted and its position will be confirmed using ultrasound guidance. Once the adequacy of the position is confirmed, the anesthesiologist will administer 15 mL of bupivacaine 0.25% with epinephrine in divided doses and examine the quality of its spread. A 20 Gauge polyamide catheter will be inserted at 2 cm in the space. The needle will then be withdrawn and the catheter will be fixed in place. Three mL of the same mixture of local anesthetics will be administered through the catheter and the anesthesiologist will observe the quality of its distribution. Bupivacaine 0.125% will be administered through the catheter using an infusion pump for 48 hours. Knee extensor muscle strength, pain and side-effects will be assessed at different time-points.
  Arms: Adductor canal femoral nerve blockade
Device: Simulated nerve blockade — The insertion of the Tuohy needle and the injection of 15 mL of bupivacaine 0.25% with epinephrine will be simulated. The insertion of the polyamide catheter, the withdrawal of the needle and the injection of local anesthetics through the catheter will also be simulated. The infusion of bupivacaine 0.125% will also be simulated for 48 hours. Knee extensor muscle strength, pain and side-effects will be assessed at different time-points.
  Arms: Simulated nerve blockade

SUMMARY:
Total knee arthroplasty (TKA) is a frequent and effective surgery for knee osteoarthritis. This major surgery is associated with a reduction in knee extensor muscle strength persisting several weeks after surgery. This decrease in strength correlates with poor functional recovery. Its cause is multifactorial, including a deficit of the quadriceps activation, an acute postoperative atrophy of the muscle and an important limitation related to postoperative pain.

Peripheral nerve blocks using local anesthetics are frequently used for postoperative analgesia following TKA. Femoral nerve blockade reduces pain and opioid consumption and allows early passive mobilization after surgery. This block also facilitates functional recovery and allows early discharge from the hospital. However, blocks involving the proximal femoral nerve contribute to quadriceps weakness for the duration of nerve blockade. Quadriceps weakness, in turn, results in functional impairment and increases recovery time. A possible long-term quadriceps weakness associated with the femoral nerve block has even been suggested in a recently published abstract. Hence, there is a need for an alternative technique that could minimize postoperative pain as well as the femoral nerve block without causing weakness of the quadriceps muscle.

Femoral nerve block performed at the level of the adductor canal seems to be a promising alternative to the classic inguinal approach of the femoral nerve block. Studies comparing femoral nerve block performed at the canal adductor level to the inguinal approach reported a similar quality of analgesia, a reduction in motor block and a better functional recovery in the early postoperative period in the canal adductor block group. The long-term effect of femoral nerve block performed at the level of the adductor canal on knee extensor strength after surgery remains to be studied.

This study will assess knee extensor muscle strength (principally quadriceps muscle) at 24h, 48h and 6 weeks following TKA in patients having a femoral nerve block at the adductor canal level compared to a simulated block.

Hypothesis: The adductor canal block will allow superior recovery of knee extensor muscle strength when compared to a simulated block at 6 weeks after total knee arthroplasty.

DETAILED DESCRIPTION:
On arrival in the operating room, patients will be randomly assigned to receive an adductor canal block under ultrasound guidance or a simulated block.

In the adductor canal block group, a 18 Gauge Tuohy needle will be inserted and its position in the adductor canal adjacent to the femoral artery will be confirmed using ultrasound guidance. Once the adequacy of the position is confirmed, the anesthesiologist will administer 15 mL of bupivacaine 0.25% with epinephrine in divided doses and examine the quality of its spread. A 20 Gauge polyamide catheter will be inserted at 2 cm in the space. The needle will then be withdrawn and the catheter will be fixed in place. Three mL of the same mixture of local anesthetics will be administered through the catheter and the anesthesiologist will observe the quality of its distribution.

In the simulated block group, the insertion of the Tuohy needle and the injection of 15 mL of bupivacaine 0.25% with epinephrine will be simulated. The insertion of the polyamide catheter, the withdrawal of the needle and the injection of local anesthetics through the catheter will also be simulated.

Surgery will be performed under spinal anesthesia. A standardized dose of bupivacaine and morphine will be administered for spinal anesthesia.

In both groups, an infusion of local anesthetics will be initiated on arrival in the recovery room and will continue for the first 48 hours. To preserve the blinding in the simulated block group, a Luer-lock connector and a 50 mL empty pouch of intravenous fluids will be affixed to the catheter to collect the infused local anesthetics. The empty pouch will be inserted under the opaque dressing. Patients in the adductor canal block will receive an infusion of bupivacaine 0.125% at 12 mL/h and patients in the simulated block group will have an infusion of the same medication but at an infusion rate of 1 mL/h. The infusion rate will be hidden from the patient. Multimodal analgesia will be used in all patients.

Patients will be asked to complete the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire before and 6 weeks following surgery.

Knee extensor muscle strength will be measured using a hand-held dynamometer pre-operatively and 24 hours, 48 hours and 6 weeks following surgery. Pain scores at rest and during strength assessment will be collected. Opioids consumption and side-effects attributable to analgesia will be recorded. Patients will be asked to rate their global satisfaction regarding the quality of analgesia 48 hours after surgery. Time to discharge will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective unilateral total knee arthroplasty
* Ability to complete the KOOS questionnaire
* American Society of Anesthesiologists (ASA) class 1-3

Exclusion Criteria:

* Contraindication to the adductor canal block (local infection, allergy to local anesthetics)
* Surgery to be performed under general anesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Knee extensor muscle strength | 6 weeks after surgery
  Will be measured using a hand-held dynamometer

SECONDARY OUTCOMES:
Knee extensor muscle strength | 24 hours and 48 hours following surgery
  Will be measured using a hand-held dynamometer
Intensity of pain at rest | Immediately prior to surgery and 24 hours,48 hours and 6 weeks following surgery
  Will be assessed using a Visual Analog Scale (VAS) from 0 to 10: 0 being no pain at all and 10 being the worst pain imaginable
Intensity of pain during extensor muscle strength assessment | Immediately prior to surgery and 24 hours,48 hours and 6 weeks following surgery
  Will be assessed using a Visual Analog Scale (VAS) from 0 to 10: 0 being no pain at all and 10 being the worst pain imaginable
Opioid consumption | 24 and 48 hours following surgery
Side-effects attributable to analgesia | 24 and 48 hours following surgery
  The presence of nausea and emesis will be recorded
Global satisfaction regarding analgesia | 48 hours following surgery
  Will be assessed using a scale from 1 to 10: 1 being totally dissatisfied and 10 being totally satisfied
Physical function in daily life | Immediately prior to surgery and 6 weeks following surgery
  Will be assessed using the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
Time to discharge from hospital | Patients will be followed for the duration of hospital stay, an average of 4 days

CONTACTS AND LOCATIONS:
Overall Officials: François Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Williams SR. In Response. Anesth Analg. 2018 Sep;127(3):e50-e51. doi: 10.1213/ANE.0000000000003571. No abstract available. PMID 29905615